CLINICAL TRIAL: NCT03740763
Title: Treatment of Neuropathic Pain With Spinal Cord Stimulation and Physiotherapy for More Effective Pain Relief, Increased Physical Activity and Improved Health Related Quality of Life
Brief Title: Spinal Cord Stimulation and Physiotherapy for Treatment of Neuropathic Pain
Acronym: SCS-PHYSIO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated prematurely due to slow inclusion rate due to the COVID-19 pandemic.
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VGRFOU-216271
Record Dates: First submitted 2018-05-09; First posted 2018-11-14 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Neuropathic Pain
Keywords: Pain; Quality of Life; Electric Stimulation Therapy; Physiotherapy
MeSH Terms: conditions — Neuralgia; Pain | interventions — Spinal Cord Stimulation; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Care Provider and Participants ar not masked. Data analysis of accelerometer data is masked (outcome assessor).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Spinal Cord Stimulation (SCS) (Active Comparator): Spinal Cord Stimulation (SCS)
  1. Pharmacological analgetic treatment and treatment with SCS for 3 months
  2. Add-on physiotherapy for 6 months to SCS and pharmacological analgetic treatment
  3. Pharmacological analgetic treatment, SCS treatment and add-on self management physical activity for 12 months
  Interventions: Device: Spinal Cord Stimulation (SCS); Other: Physiotherapy
- Physiotherapy (Active Comparator): Physiotherapy
  1. Pharmacological analgetic treatment for 3 months
  2. Physiotherapy for 3 months and pharmacological analgetic treatment
  3. Add-on SCS in combination with physiotherapy and pharmacological analgetic treatment for 3 months
  4. Pharmacological analgetic treatment, SCS treatment and add-on self management physical activity for 12 months
  Interventions: Device: Spinal Cord Stimulation (SCS); Other: Physiotherapy

INTERVENTIONS:
Device: Spinal Cord Stimulation (SCS) — SCS for treatment of neuropathic pain
Other: Physiotherapy — Physiotherapy 2 hours/week with physiotherapist and physical activity counseling for treatment of neuropathic pain

SUMMARY:
The study evaluates the combined effect of optimized pharmacological treatment, spinal cord stimulation and physiotherapy on pain relief, health-related quality of life and physical function in patients with neuropathic pain. All patients will receive optimized pharmacological treatment before start of spinal cord stimulation treatment. Half of the participants will be randomized to physiotherapy before start of spinal cord stimulation treatment while the other half will start physiotherapy after spinal cord stimulation treatment.

DETAILED DESCRIPTION:
Previous studies have indicated that almost half of the patients with moderate-severe pain receive inadequate pain relief. Neuropathic pain is a common pain condition, affecting 1.5-8% of the population. Conventional pharmacological treatment reduces pain but is often insufficient. Spinal cord stimulation (SCS) is associated with improved pain relief and health-related quality of life compared to conventional medical management. Despite SCS treatment, only half of the patients report >50% pain relief. Other studies have indicated that active, specific physiotherapy led by professionals reduces pain in chronic pain conditions. The aim of the study is to access the combined effect of optimized pharmacological treatment, SCS and physiotherapy on pain relief, health-related quality of life and physical function in patients with neuropathic pain. Furthermore, the study evaluates when it is most effective to start the physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Neuropathic pain > 6 months
* Pain intensity ≥ 5 according to NRS (for neuropathic pain component to be treated with SCS)
* Known cause of the pain
* Neuroanatomical correlation to the pain
* ≥50% of the painful area is to be treated with SCS
* The patient has a physical and psychological health status that allows the patient to participate in physiotherapy and undergo SCS implantation.

Exclusion Criteria:

* Not able to undergo SCS implantation
* Inadequate knowledge of the Swedish language
* Alcohol or substance abuse
* Severe untreated psychiatric disorders including psychiatric disease and/or psychological conditions which are the primary determinant to the patient's pain condition
* Incapacitating pain conditions of other causes than neuropathic pain
* Pregnancy
* Insufficient compliance
* Malignant disease with short expected survival

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Pain intensity according to numeric rating scale (NRS) | 3 months after implantation
  Number of patients who report ≥50% pain reduction (pain intensity) according to numeric rating scale (score from 0 to 10, where 0 is described as "no pain" and 10 as "worst pain imaginable") with regard to neuropathic pain.

SECONDARY OUTCOMES:
Pain intensity according to NRS | 9 months after implantation
  Number of patients who report ≥50% pain reduction (pain intensity) according to numeric rating scale (score from 0 to 10, where 0 is described as "no pain" and 10 as "worst pain imaginable") with regard to neuropathic pain.
Pain intensity according to NRS | 6 months after implantation
  Number of patients who report ≥50% pain reduction (pain intensity) according to numeric rating scale (score from 0 to 10, where 0 is described as "no pain" and 10 as "worst pain imaginable") with regard to neuropathic pain.
Pain intensity according to NRS | 12 months after implantation
  Number of patients who report ≥50% pain reduction (pain intensity) according to numeric rating scale (score from 0 to 10, where 0 is described as "no pain" and 10 as "worst pain imaginable") with regard to neuropathic pain.
Pain intensity according to NRS | 15 months after implantation
  Number of patients who report ≥50% pain reduction (pain intensity) according to numeric rating scale (score from 0 to 10, where 0 is described as "no pain" and 10 as "worst pain imaginable") with regard to neuropathic pain.
Pain intensity according to NRS | 21 months after implantation
  Number of patients who report ≥50% pain reduction (pain intensity) according to numeric rating scale (score from 0 to 10, where 0 is described as "no pain" and 10 as "worst pain imaginable") with regard to neuropathic pain.
Health Related Quality of Life (HRQL) according to SF36 | 3 months after implantation
  Assessed with RAND Short Form 36 (SF36). The 36 items in the questionnaire are grouped into eight subscale scores: physical functioning, role limitations caused by physical problems, bodily pain, general health, energy/vitality, social functioning, role limitations caused by emotional problems and mental health. The subscale scores range from 0-100, the higher score, the better health related quality of life.
Health Related Quality of Life (HRQL) according to SF36 | 6 months after implantation
  Assessed with RAND Short Form 36 (SF36). The 36 items in the questionnaire are grouped into eight subscale scores: physical functioning, role limitations caused by physical problems, bodily pain, general health, energy/vitality, social functioning, role limitations caused by emotional problems and mental health. The subscale scores range from 0-100, the higher score, the better health related quality of life.
Health Related Quality of Life (HRQL) according to SF36 | 9 months after implantation
  Assessed with RAND Short Form 36 (SF36). The 36 items in the questionnaire are grouped into eight subscale scores: physical functioning, role limitations caused by physical problems, bodily pain, general health, energy/vitality, social functioning, role limitations caused by emotional problems and mental health. The subscale scores range from 0-100, the higher score, the better health related quality of life.
Health Related Quality of Life (HRQL) according to SF36 | 12 months after implantation
  Assessed with RAND Short Form 36 (SF36). The 36 items in the questionnaire are grouped into eight subscale scores: physical functioning, role limitations caused by physical problems, bodily pain, general health, energy/vitality, social functioning, role limitations caused by emotional problems and mental health. The subscale scores range from 0-100, the higher score, the better health related quality of life.
Health Related Quality of Life (HRQL) according to SF36 | 15 months after implantation
  Assessed with RAND Short Form 36 (SF36). The 36 items in the questionnaire are grouped into eight subscale scores: physical functioning, role limitations caused by physical problems, bodily pain, general health, energy/vitality, social functioning, role limitations caused by emotional problems and mental health. The subscale scores range from 0-100, the higher score, the better health related quality of life.
Health Related Quality of Life (HRQL) according to SF36 | 21 months after implantation
  Assessed with RAND Short Form 36 (SF36). The 36 items in the questionnaire are grouped into eight subscale scores: physical functioning, role limitations caused by physical problems, bodily pain, general health, energy/vitality, social functioning, role limitations caused by emotional problems and mental health. The subscale scores range from 0-100, the higher score, the better health related quality of life.
Health Related Quality of Life (HRQL) assessed with EQ-5D | 3 months after implantation
  Assessed with EQ-5D-5L. The questionnaire comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Health Related Quality of Life (HRQL) assessed with EQ-5D | 6 months after implantation
  Assessed with EQ-5D-5L. The questionnaire comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Health Related Quality of Life (HRQL) assessed with EQ-5D | 9 months after implantation
  Assessed with EQ-5D-5L. The questionnaire comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Health Related Quality of Life (HRQL) assessed with EQ-5D | 12 months after implantation
  Assessed with EQ-5D-5L. The questionnaire comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Health Related Quality of Life (HRQL) assessed with EQ-5D | 15 months after implantation
  Assessed with EQ-5D-5L. The questionnaire comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Health Related Quality of Life (HRQL) assessed with EQ-5D | 21 months after implantation
  Assessed with EQ-5D-5L. The questionnaire comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Physical activity | 3 months
  Assessed with accelerometer
Physical activity | 6 months
  Assessed with accelerometer
Physical activity | 9 months
  Assessed with accelerometer
Physical activity | 12 months
  Assessed with accelerometer
Physical activity | 15 months
  Assessed with accelerometer
Physical activity | 21 months
  Assessed with accelerometer
Return to work | 9 months
  Number of patients who return to work part time or full time.
Return to work | 21 months
  Number of patients who return to work part time or full time.
Days of sick-leave | 9 months
  Number of days of sick-leave
Days of sick-leave | 21 months
  Number of days of sick-leave
Medicine consumption | 9 months
  Number of pills and dosage.
Medicine consumption | 21 months
  Number of pills and dosage.
Number of hospital and primary care visits | 9 months
  Number of hospital and primary care visits
Number of hospital and primary care visits | 21 months
  Number of hospital and primary care visits
Patient treatment satisfaction according to NRS | 3 months after implantation
  Self-reported treatment satisfaction with regard to pain relief, how acceptable the patient finds the treatment and hospital care. Numeric rating scale (score from 0 to 10, where 0 is described as "not satisfied at all" and 10 as "very satisfied") and numeric rating scale (score from 0 to 10, where 0 is described as "not acceptable at all" and 10 as "very acceptable").
Patient treatment satisfaction according to NRS | 6 months after implantation
  Self-reported treatment satisfaction with regard to pain relief, how acceptable the patient finds the treatment and hospital care. Numeric rating scale (score from 0 to 10, where 0 is described as "not satisfied at all" and 10 as "very satisfied") and numeric rating scale (score from 0 to 10, where 0 is described as "not acceptable at all" and 10 as "very acceptable").
Patient treatment satisfaction according to NRS | 9 months after implantation
  Self-reported treatment satisfaction with regard to pain relief, how acceptable the patient finds the treatment and hospital care. Numeric rating scale (score from 0 to 10, where 0 is described as "not satisfied at all" and 10 as "very satisfied") and numeric rating scale (score from 0 to 10, where 0 is described as "not acceptable at all" and 10 as "very acceptable").
Patient treatment satisfaction according to NRS | 12 months after implantation
  Self-reported treatment satisfaction with regard to pain relief, how acceptable the patient finds the treatment and hospital care. Numeric rating scale (score from 0 to 10, where 0 is described as "not satisfied at all" and 10 as "very satisfied") and numeric rating scale (score from 0 to 10, where 0 is described as "not acceptable at all" and 10 as "very acceptable").
Patient treatment satisfaction according to NRS | 15 months after implantation
  Self-reported treatment satisfaction with regard to pain relief, how acceptable the patient finds the treatment and hospital care. Numeric rating scale (score from 0 to 10, where 0 is described as "not satisfied at all" and 10 as "very satisfied") and numeric rating scale (score from 0 to 10, where 0 is described as "not acceptable at all" and 10 as "very acceptable").
Patient treatment satisfaction according to NRS | 21 months after implantation
  Self-reported treatment satisfaction with regard to pain relief, how acceptable the patient finds the treatment and hospital care. Numeric rating scale (score from 0 to 10, where 0 is described as "not satisfied at all" and 10 as "very satisfied") and numeric rating scale (score from 0 to 10, where 0 is described as "not acceptable at all" and 10 as "very acceptable").

OTHER OUTCOMES:
Anxiety, depression | 3 months after implantation
  Assessed with the Hospital Anxiety and Depression (HAD) scale. The scale consists of 14 items on a four-point response scale ranging from 0-3. Seven items for depression and 7 items for anxiety with a score range from 0-21. For each factor (anxiety or depression), the results are interpreted as follows: < 8 points indicates within normal range, 8-10 points indicates possible and >10 points indicates probable anxiety or depression.
Anxiety, depression | 6 months after implantation
  Assessed with the Hospital Anxiety and Depression (HAD) scale. The scale consists of 14 items on a four-point response scale ranging from 0-3. Seven items for depression and 7 items for anxiety with a score range from 0-21. For each factor (anxiety or depression), the results are interpreted as follows: < 8 points indicates within normal range, 8-10 points indicates possible and >10 points indicates probable anxiety or depression.
Anxiety, depression | 9 months after implantation
  Assessed with the Hospital Anxiety and Depression (HAD) scale. The scale consists of 14 items on a four-point response scale ranging from 0-3. Seven items for depression and 7 items for anxiety with a score range from 0-21. For each factor (anxiety or depression), the results are interpreted as follows: < 8 points indicates within normal range, 8-10 points indicates possible and >10 points indicates probable anxiety or depression.
Anxiety, depression | 12 months after implantation
  Assessed with the Hospital Anxiety and Depression (HAD) scale. The scale consists of 14 items on a four-point response scale ranging from 0-3. Seven items for depression and 7 items for anxiety with a score range from 0-21. For each factor (anxiety or depression), the results are interpreted as follows: < 8 points indicates within normal range, 8-10 points indicates possible and >10 points indicates probable anxiety or depression.
Anxiety, depression | 15 months after implantation
  Assessed with the Hospital Anxiety and Depression (HAD) scale. The scale consists of 14 items on a four-point response scale ranging from 0-3. Seven items for depression and 7 items for anxiety with a score range from 0-21. For each factor (anxiety or depression), the results are interpreted as follows: < 8 points indicates within normal range, 8-10 points indicates possible and >10 points indicates probable anxiety or depression.
Anxiety, depression | 21 months after implantation
  Assessed with the Hospital Anxiety and Depression (HAD) scale. The scale consists of 14 items on a four-point response scale ranging from 0-3. Seven items for depression and 7 items for anxiety with a score range from 0-21. For each factor (anxiety or depression), the results are interpreted as follows: < 8 points indicates within normal range, 8-10 points indicates possible and >10 points indicates probable anxiety or depression.
Physical activity | 3 months after implantations
  Assessed with the "Saltin-Grimby Physical Activity Level Scale" (SGPALS) is a scale that measures physical activity during the last year using the question "How much do you move and exert yourself physically during your leisure time?". The question has four options, where 1 is physically inactive and 4 is regular hard physical training for competitive sports.
Physical activity | 6 months after implantations
  Assessed with the "Saltin-Grimby Physical Activity Level Scale" (SGPALS) is a scale that measures physical activity during the last year using the question "How much do you move and exert yourself physically during your leisure time?". The question has four options, where 1 is physically inactive and 4 is regular hard physical training for competitive sports.
Physical activity | 9 months after implantations
  Assessed with the "Saltin-Grimby Physical Activity Level Scale" (SGPALS) is a scale that measures physical activity during the last year using the question "How much do you move and exert yourself physically during your leisure time?". The question has four options, where 1 is physically inactive and 4 is regular hard physical training for competitive sports.
Physical activity | 12 months after implantations
  Assessed with the "Saltin-Grimby Physical Activity Level Scale" (SGPALS) is a scale that measures physical activity during the last year using the question "How much do you move and exert yourself physically during your leisure time?". The question has four options, where 1 is physically inactive and 4 is regular hard physical training for competitive sports.
Physical activity | 15 months after implantations
  Assessed with the "Saltin-Grimby Physical Activity Level Scale" (SGPALS) is a scale that measures physical activity during the last year using the question "How much do you move and exert yourself physically during your leisure time?". The question has four options, where 1 is physically inactive and 4 is regular hard physical training for competitive sports.
Physical activity | 21 months after implantations
  Assessed with the "Saltin-Grimby Physical Activity Level Scale" (SGPALS) is a scale that measures physical activity during the last year using the question "How much do you move and exert yourself physically during your leisure time?". The question has four options, where 1 is physically inactive and 4 is regular hard physical training for competitive sports.
Sleep quality according to Pittsburgh Sleep Quality Index | 3 months after implantation
  Assessed with the Pittsburgh Sleep Quality Index (PSQI). The PSQI consists of 19 self-rated questions which assess a wide variety of factors relating to sleep quality, including estimates of sleep duration and latency and of the frequency and severity of specific sleep related problems. The 19 items are grouped into seven component scores, each weighted equally on a 0-3 scale. The seven component score are then summed to yield a global PSQI score which has a range of 0-21; higher scores indicate worse sleep quality.
Sleep quality according to Pittsburgh Sleep Quality Index | 6 months after implantation
  Assessed with the Pittsburgh Sleep Quality Index (PSQI). The PSQI consists of 19 self-rated questions which assess a wide variety of factors relating to sleep quality, including estimates of sleep duration and latency and of the frequency and severity of specific sleep related problems. The 19 items are grouped into seven component scores, each weighted equally on a 0-3 scale. The seven component score are then summed to yield a global PSQI score which has a range of 0-21; higher scores indicate worse sleep quality.
Sleep quality according to Pittsburgh Sleep Quality Index | 9 months after implantation
  Assessed with the Pittsburgh Sleep Quality Index (PSQI). The PSQI consists of 19 self-rated questions which assess a wide variety of factors relating to sleep quality, including estimates of sleep duration and latency and of the frequency and severity of specific sleep related problems. The 19 items are grouped into seven component scores, each weighted equally on a 0-3 scale. The seven component score are then summed to yield a global PSQI score which has a range of 0-21; higher scores indicate worse sleep quality.
Sleep quality according to Pittsburgh Sleep Quality Index | 12 months after implantation
  Assessed with the Pittsburgh Sleep Quality Index (PSQI). The PSQI consists of 19 self-rated questions which assess a wide variety of factors relating to sleep quality, including estimates of sleep duration and latency and of the frequency and severity of specific sleep related problems. The 19 items are grouped into seven component scores, each weighted equally on a 0-3 scale. The seven component score are then summed to yield a global PSQI score which has a range of 0-21; higher scores indicate worse sleep quality.
Sleep quality according to Pittsburgh Sleep Quality Index | 15 months after implantation
  Assessed with the Pittsburgh Sleep Quality Index (PSQI). The PSQI consists of 19 self-rated questions which assess a wide variety of factors relating to sleep quality, including estimates of sleep duration and latency and of the frequency and severity of specific sleep related problems. The 19 items are grouped into seven component scores, each weighted equally on a 0-3 scale. The seven component score are then summed to yield a global PSQI score which has a range of 0-21; higher scores indicate worse sleep quality.
Sleep quality according to Pittsburgh Sleep Quality Index | 21 months after implantation
  Assessed with the Pittsburgh Sleep Quality Index (PSQI). The PSQI consists of 19 self-rated questions which assess a wide variety of factors relating to sleep quality, including estimates of sleep duration and latency and of the frequency and severity of specific sleep related problems. The 19 items are grouped into seven component scores, each weighted equally on a 0-3 scale. The seven component score are then summed to yield a global PSQI score which has a range of 0-21; higher scores indicate worse sleep quality.
Kinesiophobia | 3 months
  Assessed with Tampa Scale of Kinesiophobia (TSK). The TSK is a 17 item scale, developed to measure pain related fear of movement. A total scores from 17 to 68 is calculated where the higher scores indicate an increasing degree of kinesiophobia.
Kinesiophobia | 6 months
  Assessed with Tampa Scale of Kinesiophobia (TSK). The TSK is a 17 item scale, developed to measure pain related fear of movement. A total scores from 17 to 68 is calculated where the higher scores indicate an increasing degree of kinesiophobia.
Kinesiophobia | 9 months
  Assessed with Tampa Scale of Kinesiophobia (TSK). The TSK is a 17 item scale, developed to measure pain related fear of movement. A total scores from 17 to 68 is calculated where the higher scores indicate an increasing degree of kinesiophobia.
Kinesiophobia | 12 months
  Assessed with Tampa Scale of Kinesiophobia (TSK). The TSK is a 17 item scale, developed to measure pain related fear of movement. A total scores from 17 to 68 is calculated where the higher scores indicate an increasing degree of kinesiophobia.
Kinesiophobia | 15 months
  Assessed with Tampa Scale of Kinesiophobia (TSK). The TSK is a 17 item scale, developed to measure pain related fear of movement. A total scores from 17 to 68 is calculated where the higher scores indicate an increasing degree of kinesiophobia.
Kinesiophobia | 21 months
  Assessed with Tampa Scale of Kinesiophobia (TSK). The TSK is a 17 item scale, developed to measure pain related fear of movement. A total scores from 17 to 68 is calculated where the higher scores indicate an increasing degree of kinesiophobia.
Self-efficacy: A-SES-S | 3 months
  Assessed with self-efficacy for arthritis (A-SES-S). A-SES is a self-efficacy questionnaire that contains 20 questions and measure a paitent's self-efficacy in three categories: capacity to handle pain, function and other symptoms. A total score between 10 and 100 is calculated, were a high total score indicates a high self-efficacy. The three categories can also be calculated separately and divided in number of questions also resulting of a score between 10 and 100. In the study we will analyze the categories "capacity to handle pain" and "other symptoms".
Self-efficacy: A-SES-S | 6 months
  Assessed with self-efficacy for arthritis (A-SES-S). A-SES is a self-efficacy questionnaire that contains 20 questions and measure a paitent's self-efficacy in three categories: capacity to handle pain, function and other symptoms. A total score between 10 and 100 is calculated, were a high total score indicates a high self-efficacy. The three categories can also be calculated separately and divided in number of questions also resulting of a score between 10 and 100. In the study we will analyze the categories "capacity to handle pain" and "other symptoms".
Self-efficacy | 9 months
  Assessed with self-efficacy for arthritis (A-SES-S). A-SES is a self-efficacy questionnaire that contains 20 questions and measure a paitent's self-efficacy in three categories: capacity to handle pain, function and other symptoms. A total score between 10 and 100 is calculated, were a high total score indicates a high self-efficacy. The three categories can also be calculated separately and divided in number of questions also resulting of a score between 10 and 100. In the study we will analyze the categories "capacity to handle pain" and "other symptoms".
Self-efficacy: A-SES-S | 12 months
  Assessed with self-efficacy for arthritis (A-SES-S). A-SES is a self-efficacy questionnaire that contains 20 questions and measure a paitent's self-efficacy in three categories: capacity to handle pain, function and other symptoms. A total score between 10 and 100 is calculated, were a high total score indicates a high self-efficacy. The three categories can also be calculated separately and divided in number of questions also resulting of a score between 10 and 100. In the study we will analyze the categories "capacity to handle pain" and "other symptoms".
Self-efficacy: A-SES-S | 15 months
  Assessed with self-efficacy for arthritis (A-SES-S). A-SES is a self-efficacy questionnaire that contains 20 questions and measure a paitent's self-efficacy in three categories: capacity to handle pain, function and other symptoms. A total score between 10 and 100 is calculated, were a high total score indicates a high self-efficacy. The three categories can also be calculated separately and divided in number of questions also resulting of a score between 10 and 100. In the study we will analyze the categories "capacity to handle pain" and "other symptoms".
Self-efficacy: A-SES-S | 21 months
  Assessed with self-efficacy for arthritis (A-SES-S). A-SES is a self-efficacy questionnaire that contains 20 questions and measure a paitent's self-efficacy in three categories: capacity to handle pain, function and other symptoms. A total score between 10 and 100 is calculated, were a high total score indicates a high self-efficacy. The three categories can also be calculated separately and divided in number of questions also resulting of a score between 10 and 100. In the study we will analyze the categories "capacity to handle pain" and "other symptoms".
Self-efficacy for exercise | 3 months
  Assessed with self-efficacy for exercise (SEE-SV). The self efficacy scale measures a patient's self-efficacy when it comes to physical exercise. The questionnaire consists of 9 questions that can be answered on a 1-10 scale. A total score between 9 and 90 is calculated, were a higher number represent a better outcome.
Self-efficacy for exercise | 6 months
  Assessed with self-efficacy for exercise (SEE-SV). The self efficacy scale measures a patient's self-efficacy when it comes to physical exercise. The questionnaire consists of 9 questions that can be answered on a 1-10 scale. A total score between 9 and 90 is calculated, were a higher number represent a better outcome.
Self-efficacy for exercise | 9 months
  Assessed with self-efficacy for exercise (SEE-SV). The self efficacy scale measures a patient's self-efficacy when it comes to physical exercise. The questionnaire consists of 9 questions that can be answered on a 1-10 scale. A total score between 9 and 90 is calculated, were a higher number represent a better outcome.
Self-efficacy for exercise | 12 months
  Assessed with self-efficacy for exercise (SEE-SV). The self efficacy scale measures a patient's self-efficacy when it comes to physical exercise. The questionnaire consists of 9 questions that can be answered on a 1-10 scale. A total score between 9 and 90 is calculated, were a higher number represent a better outcome.
Self-efficacy for exercise | 15 months
  Assessed with self-efficacy for exercise (SEE-SV). The self efficacy scale measures a patient's self-efficacy when it comes to physical exercise. The questionnaire consists of 9 questions that can be answered on a 1-10 scale. A total score between 9 and 90 is calculated, were a higher number represent a better outcome.
Self-efficacy for exercise | 21 months
  Assessed with self-efficacy for exercise (SEE-SV). The self efficacy scale measures a patient's self-efficacy when it comes to physical exercise. The questionnaire consists of 9 questions that can be answered on a 1-10 scale. A total score between 9 and 90 is calculated, were a higher number represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Paulin Andréll, MD, PhD, Principal Investigator — Göteborgs Universitet/Västra Götalandsregionen
Locations (1):
- Pain center, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gottfridsson R, Varkey E, Wolf A, Gatzinsky K, Liljencrantz J, Thorn SE, Borjesson M, Arvidsson D, Andrell P. Effects of spinal cord stimulation on pain, physical activity, and self-efficacy among patients with neuropathic pain. Pain Manag. 2026 Jan 7:1-15. doi: 10.1080/17581869.2025.2608572. Online ahead of print. PMID 41503863
- [Derived] O'Connell NE, Ferraro MC, Gibson W, Rice AS, Vase L, Coyle D, Eccleston C. Implanted spinal neuromodulation interventions for chronic pain in adults. Cochrane Database Syst Rev. 2021 Dec 2;12(12):CD013756. doi: 10.1002/14651858.CD013756.pub2. PMID 34854473
- See also: Project description in Swedish — https://www.researchweb.org/is/vgr/project/216271